Principal Investigator: Virginia Sun, PhD, RN

Department/Division: Population Sciences, Division of Nursing Research and Education

Telephone number: 626-218-3122



## ADDENDUM TO INFORMED CONSENT FOR PARTICIPATION IN RESEARCH ACTIVITIES IRB#17238 - A Multimedia Self-Management Intervention to Prepare Family Caregivers and Patients for Lung Cancer Surgery

## PATIENT VERSION

Addendum [a, etc.]: [Social Determinants of Health]

<u>PURPOSE OF THIS ADDENDUM CONSENT FORM</u>: Previously you signed an informed consent form before you became a research participant in the above study. In that consent form, you were told that you would be informed of any new information that might affect your willingness to continue to participate. The purpose of this Addendum to Informed Consent is to advise you of the following new information.

You will be asked to complete an additional questionnaire about how your living environment, neighborhood, social support networks, and employment impacts your cancer care. You will also be asked to complete an additional questionnaire on your spiritual well-being. You will complete these questionnaires when you agree to join the study. Questionnaires can be completed in person, or by phone, or electronically via internet.

## **INFORMED CONSENT**

IRB NUMBER: 17238

IRB APPROVED FROM: 04/07/2023 IRB APPROVED TO: 04/06/2024 Name:

DOB :

MRN#:

FORM NO 8700-C037 09/28/2021

| original consent form that you signed remain in effe | | |
|---|---|---|
| Research Participant's Signature | Date | Time |
| (For paper consent only, then the date and tin | me must be in research | participant's handwriting) |
| Print Research Participant's Name | | |
| Tint Research Participant's Name | | |
| INDIVIDUAL OBTAINING CONSENT SIGNA | TURE | |
| Signature of Individual Obtaining Consent | Date | Time |
| Signature of Individual Obtaining Consent | Date | Time |
| | Date | Time |
| Print Name of Individual Obtaining Consent Originature of Individual Obtaining Consent | Date | Time |
| | Date | Time |
| | Date | Time |
| | Date | Time |
| | Date | Time |

## **INFORMED CONSENT**

IRB NUMBER: 17238

IRB APPROVED FROM: 04/07/2023 IRB APPROVED TO: 04/06/2024 Name :

DOB :

MRN#: